CLINICAL TRIAL: NCT05203744
Title: Safety, Tolerability and Pharmacokinetics of Tafenoquine After Weekly and Escalating Monthly Doses of Tafenoquine in Healthy Vietnamese Volunteers
Brief Title: Escalating Monthly Doses of Tafenoquine in Healthy Volunteers
Acronym: TQ
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Naval Medical Research Center (U.S. Federal Agency)
Collaborators: Naval Medical Research Unit TWO (NAMRU-2) (Unknown); Australian Defence Force Malaria and Infectious Disease Institute (ADF MIDI) (Unknown); The 108 Military Central Hospital (Other Government); Naval Environmental Preventive Medicine Unit TWO (NEPMU-2) (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Prevention
Other Study IDs: NAMRU2.2021.0002
Record Dates: First submitted 2021-12-20; First posted 2022-01-24 (Actual); Last update posted 2022-04-11 (Actual); Status verified 2022-04

CONDITIONS: Prophylaxis
Keywords: malaria; prophylaxis; tafenoquine; Vietnam
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Intervention Model Description: The 200 healthy participants will be divided into two cohorts (A and B) of 100 participants to fully cover the three tafenoquine regimens (i.e. weekly, low monthly and high monthly) in obtaining study information (e.g. AEs) and biospecimens for monitoring the safety, tolerability and PK of tafenoquine.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Standard Dose (200 mg) (Experimental): Participants will receive the standard 200 mg tafenoquine dose (200 mg daily for 3 days) followed by 200 mg weekly for two weeks to check for tolerability and adverse effects.
  Interventions: Drug: Tafenoquine prophylaxis
- Low Monthly Dose (600 mg) (Experimental): The same participants from Part 1 will be administered a monthly dose of tafenoquine (600 mg total, given as 300 mg split over 2 days) for two consecutive months. This monthly dose of 600 mg tafenoquine is designated the "low" monthly tafenoquine dose.
  Interventions: Drug: Tafenoquine prophylaxis
- High Monthly Dose (800 mg) (Experimental): The same participants from Parts 1 and 2 will be administered a monthly dose of tafenoquine (800 mg total, given as 400 mg split over 2 days) for two consecutive months. This monthly dose of 800 mg tafenoquine is designated the high monthly tafenoquine dose
  Interventions: Drug: Tafenoquine prophylaxis

INTERVENTIONS:
Drug: Tafenoquine prophylaxis — The study will be conducted in three parts with 200 participants invited to participate in the study.
  * Part 1 consist of 200 participants to be administered a loading dose of 600 mg tafenoquine (200 mg daily for 3 days) followed by 200 mg weekly for two weeks.
  * Part 2: The same participants from Part 1 will be administered a monthly dose of tafenoquine (600 mg total, given as 300 mg split over 2 days) for two consecutive months. This monthly dose of 600 mg tafenoquine is designated the "low" monthly tafenoquine dose.
  * Part 3: The same participants from Parts 1 and 2 will be administered a monthly dose of tafenoquine (800 mg total, given as 400 mg split over 2 days) for two consecutive months. This monthly dose of 800 mg tafenoquine is designated the high monthly tafenoquine dose.
  Other Names: TQ

SUMMARY:
In 2018, the U.S. Food and Drug Administration (FDA) and the Australian Therapeutic Goods Administration (TGA) approved tafenoquine for malaria prevention. The approved tafenoquine prophylactic regimen is 600 mg loading dose (200 mg daily for 3 days) prior to travel and a weekly 200 mg maintenance dose commencing 7 days after the last loading dose. This weekly tafenoquine regimen is more convenient with potentially improved compliance than daily doxycycline or atovaquone proguanil (Malarone), the other recommended prophylactic agents by the U.S. Centers for Disease Control and Prevention (CDC) for the prevention of malaria infections.

Current assumptions are that a systemic minimum inhibitory concentration (MIC) of tafenoquine in plasma is 80 ng/mL in nonimmune individuals is required to prevent symptomatic breakthroughs of malaria infections. Because of tafenoquine's lengthy blood elimination half-life of 2-3 weeks, a monthly regimen of 600 mg and 800 mg of tafenoquine in individuals weighing 60 kg and 80 kg, respectively, have pharmacokinetic (PK) profiles (i.e., drug concentration versus time curves) of achieving MIC values of at least 80 ng/mL in the majority of healthy individuals. The aim of this study is to determine whether the safety and tolerability profiles in healthy participants taking monthly doses of 600 mg or 800 mg tafenoquine are comparable in the same participants taking weekly 200 mg tafenoquine.

Study Hypothesis: The study hypothesis is that the frequency of tafenoquine-related safety (e.g. blood chemistries) and adverse events (AEs) in healthy participants who take a higher dose (600 mg and 800 mg) of tafenoquine monthly would be comparable to the frequency of treatment related safety and AEs in the same individuals who take weekly tafenoquine (200 mg).

DETAILED DESCRIPTION:
This is an open-label study to evaluate the safety, tolerability and PK of tafenoquine after weekly and two monthly doses of tafenoquine in healthy participants. The study will be conducted in three parts with 200 participants invited to participate in the study.

* Part 1 consist of 200 participants to be administered a loading dose of 600 mg tafenoquine (200 mg daily for 3 days) followed by 200 mg weekly for two weeks.
* Part 2: The same participants from Part 1 will be administered a monthly dose of tafenoquine (600 mg total, given as 300 mg split over 2 days) for two consecutive months. This monthly dose of 600 mg tafenoquine is designated the "low" monthly tafenoquine dose.
* Part 3: The same participants from Parts 1 and 2 will be administered a monthly dose of tafenoquine (800 mg total, given as 400 mg split over 2 days) for two consecutive months. This monthly dose of 800 mg tafenoquine is designated the high monthly tafenoquine dose.

The 200 healthy participants will be divided into two cohorts (A and B) of 100 participants to fully cover the three tafenoquine regimens (i.e. weekly, low monthly and high monthly) in obtaining study information (e.g. AEs) and biospecimens for monitoring the safety, tolerability and PK of tafenoquine.

Tafenoquine: Arakoda™ tablets (each containing 100 mg of tafenoquine base) are dark pink, capsule shaped, debossed with "TQ100" on one side and plain on the other. Arakoda™ tablets are supplied in blister packs. Each blister pack contains 8 tablets. Monthly tafenoquine will be administered as 100 mg oral tafenoquine tablets (Arakoda™) identical to those marketed for weekly prophylaxis.

Objectives: Primary Objective: In a dose escalating study in the same healthy participants compare the frequency of treatment-related safety and adverse events (AEs) after weekly 200 mg tafenoquine and two monthly (600 mg and 800 mg) tafenoquine regimens.

Secondary Objectives:

* Characterize the PK profiles of tafenoquine after weekly 200 mg and two monthly (600 mg and 800 mg) tafenoquine regimens in the same healthy participants.
* Characterize the pharmacokinetic/pharmacodynamic (PK/PD) relationship between blood tafenoquine concentrations and safety and tolerability of the weekly 200 mg and two monthly (600 mg or 800 mg) tafenoquine regimens in the same healthy participants.
* Determine the association of tafenoquine and its metabolite 5,6, orthoquinone in red blood cells, the site of action of the drug's blood schizontocidal activity.
* Determine the ex vivo antimalarial activity of tafenoquine in participants' plasma samples after tafenoquine administration (weekly and monthly regimens) against Plasmodium falciparum strains with different levels of drug susceptibility.

Study Population: Two hundred healthy participants are planned to be enrolled in this study for Parts 1 to 3. It is planned to recruit 200 participants from 108 Military Central Hospital.

The healthy participants will be judged to be in good health based on medical history, physical examination, blood chemistries, urinalysis, serology, normal electrocardiogram (ECG), glucose-6-phosphate dehydrogenase (G6PD) normal, and free of infectious diseases, psychiatric concerns, allergies and other medical conditions that the Investigator deems may compromise the potential participant's safety and wellbeing.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female aged 18 to 55 years inclusive who will be contactable and available for the duration of the study.
2. Total body weight greater than or equal to 45 kg, and a body mass index (BMI) within the range of 18 to 32 kg/m2 (inclusive).
3. Vietnamese (Kinh people) or belonging to one of the other 53 ethnic groups in Vietnam.
4. G6PD enzyme activity levels of >70% of the site median value for normal G6PD using a quantitative G6PD test.
5. Certified as in good health as determined by a comprehensive clinical assessment (past medical history, complete physical examination, vital signs, ECG) and laboratory tests (biochemical, hematology and urinalysis results at screening that are within the local laboratory reference range).
6. Vital signs at screening and throughout the study (measured after five minutes in the supine position) within the following ranges:

   * Systolic blood pressure (SBP) - 90-140 mmHg.
   * Diastolic blood pressure (DBP) - 40-90 mmHg.
   * Heart rate (HR) 40-100 bpm.
7. ECG ranges at screening: Time from the start of the Q wave to the end of the T wave (QT) corrected (QTc) by Bazett's formula (QTcB)/QT interval corrected by Fridericia's formula (QTcF) ≤450 ms for male participants, QTcB/QTcF ≤470 ms for female participants, and Pulse Rate (PR) interval ≤210 ms.
8. A female participant of childbearing potential is eligible to enter the study if she is non-pregnant, non-lactating, has a negative pregnancy test at the screening visit and agrees to comply with one of the following contraceptive procedures during the study and for a period of 90 days after the last dose of tafenoquine.

   - Use of oral contraceptive, either combined or progestogen alone used in conjunction with a double barrier method.

   - Use of an intrauterine device with a documented failure rate of <1% per year.

   - Use of depo provera injection.

   - Double barrier method consisting of spermicide with either condom or diaphragm.

   - Male partner who is sterile prior to the female participant's entry into the study and is the sole sexual partner for the female.

   - Complete abstinence from intercourse for two weeks prior to tafenoquine administration, throughout the study and for a period of 90 days after the last dose of tafenoquine.
9. Women of non-childbearing potential who will not require contraception during the study are defined as: surgically sterile or post-menopausal.
10. Male participants who have, or may have, female sexual partner(s) during the course of the study must agree to one of the following acceptable double methods of contraception:

    - Condom plus diaphragm or condom plus insertable device, or condom plus stable oral/transdermal/injectable hormonal contraceptive by the female partner.

    - Surgical sterilization (vasectomy) and a barrier method (condom or occlusive cap).
11. Abstinent male participants must agree to start a double method of contraception if they begin sexual relationships with a female during the study.
12. Willing and able to comply with all scheduled visits, physical examination, AE questionnaire, laboratory tests, and other study procedures.
13. Willingness to complete an acceptability questionnaire after each tafenoquine regimen.
14. Completion of the written informed consent process prior to undertaking any study-related procedure.

Exclusion Criteria:

1. Female participants who are pregnant or breast feeding (lactating).
2. Resting vital signs (measured after 5 minutes) at screening outside of the following ranges:

   * Body temperature (i.e. tympanic body temperature >38.0°C).
   * 40 ≤ PR ≥ 100 bpm.
   * 90 ≤ SBP ≥ 140 mmHg.
   * 50 ≤ DBP ≥ 90 mmHg.
3. Presence of acute infectious disease or fever (i.e. tympanic body temperature >38.0°C) within 5 days prior to the first dose of study medication.
4. Cardiac/QT risk:

   - Family history of sudden death or of congenital prolongation of the QTc interval or known congenital prolongation of the QTc interval or any clinical condition known to prolong the QTc interval.
   * History of symptomatic cardiac arrhythmias or with clinically relevant bradycardia.
   * Electrolyte disturbances, particularly hypokalemia, hypocalcaemia, or hypomagnesaemia.
   * ECG abnormalities in the standard 12-lead ECG at screening which in the opinion of the PI/Co-PI is clinically relevant or will interfere with the ECG analyses.
5. Positive result for any of the following serology tests: hepatitis B surface antigen (HBs Ag), anti-hepatitis B core antibodies (anti-HBc Ab), anti-hepatitis C virus (anti-HCV) antibodies, anti-human immunodeficiency virus 1 and 2 antibodies (anti-HIV1 and anti-HIV2 Ab).
6. Any recent (<6 weeks) or current systemic therapy with an antibiotic or drug with potential antimalarial activity (e.g. azithromycin, clindamycin, doxycycline, trimethoprim/sulfamethoxazole, hydroxychloroquine etc.) (only participants providing blood for ex vivo antimalarial studies of tafenoquine).
7. Participants are currently taking medications and chemicals that are commonly associated with the development of hemolytic anemia such as chloroquine, dapsone, fava beans, flutamide, methylthioninium chloride, nitrofurantoin, pegloticase, phenazopyridine, primaquine, rasburicase, and trimethoprim/sulfamethoxazole.
8. History or presence of diagnosed (by an allergist/immunologist) or treated (by a physician) food or known drug allergies or any history of anaphylaxis or other severe allergic reactions including face, mouth, or throat swelling or any difficulty breathing. Participants with seasonal allergies/hay fever can be enrolled in the study.
9. Presence of current or suspected serious chronic diseases such as cardiac or autoimmune disease, insulin-dependent and non-insulin dependent diabetes, progressive neurological disease, severe malnutrition, acute or progressive hepatic disease, acute or progressive renal disease, porphyria, psoriasis, rheumatoid arthritis, asthma (excluding childhood asthma, or mild asthma with preventative asthma medication required less than monthly), epilepsy, or obsessive-compulsive disorder.
10. History of malignancy of any organ system (other than localized basal cell carcinoma of the skin or in situ cervical cancer), treated or untreated, within five years of screening, regardless of whether there is evidence of local recurrence or metastases.
11. Participants with history of schizophrenia, bi-polar disease, psychoses, disorders requiring lithium, attempted or planned suicide, or any other severe (disabling) chronic psychiatric diagnosis.
12. Participants who have received psychiatric medications within one year prior to screening, or who have been hospitalized within five years prior to screening for either a psychiatric illness or due to danger to self or others.
13. History of an episode of minor depression that required at least six months of pharmacological therapy and/or psychotherapy within the last five years; or any episode of major depression. The Beck Depression Inventory (BDI) will be used as an objective tool for the assessment of depression at screening.

4. History of recurrent headache (e.g. tension-type, cluster or migraine), recurrent nausea, and/or vomiting with a frequency of ≥2 episodes per month on average and severe enough to require medical therapy, during the six months preceding the screening visit.

15. Evidence of acute illness within the four weeks prior to screening that the PI/Co-investigator deems may compromise participant safety.

16. Significant inter-current disease of any type, in particular liver, renal, cardiac, pulmonary, neurologic, rheumatologic, or autoimmune disease by history, physical examination, and/or laboratory studies including urinalysis.

17. Participant has a clinically significant disease or any condition or disease that might affect drug absorption, distribution or excretion (e.g. gastrectomy, diarrhea).

18. Use of prescription or non-prescription drugs, herbal and dietary supplements within 14 days or five blood elimination half-lives (whichever is the longer) prior to the first dose of tafenoquine. The exceptions are: Ibuprofen (preferred) may be used at doses of up to 1.2 g per day or paracetamol at doses of up to 4 g per day. Limited use of other non-prescription medications or dietary supplements not believed to affect participant safety or the overall results of the study may be permitted on a case-by-case basis following approval by the Sponsor in consultation with the PI or Co-investigator.

19. History of retinal abnormalities, diseases of the retina or macula of the eye, visual field defects, and hearing disorders like reduced hearing and tinnitus.

20. Any participant who, in the judgment of the PI or Co-investigator, is likely to be non-compliant during the study, or is unable to cooperate because of a language problem or poor mental development.

21. Any participant who is directly involved in conducting the study. 22. Any participant with poor peripheral venous access for blood sampling. 23. Known hypersensitivity reactions to primaquine, other 8-aminoquinolines, or any component of Arakoda™.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Estimated)
Dates: Start 2022-05-10 (Estimated); Primary Completion 2022-12-03 (Estimated); Study Completion 2022-12-03 (Estimated)

PRIMARY OUTCOMES:
Tafenoquine dose escalating study to compare the frequency of treatment-related safety and adverse events and minimum inhibitory concentration of the medication after weekly 200 mg tafenoquine and two monthly (600 mg and 800 mg) tafenoquine regimens. | six months
  In a dose escalating study in the same healthy participants compare the frequency of treatment-related safety and adverse events (AEs) after weekly 200 mg tafenoquine and two monthly (600 mg and 800 mg) tafenoquine regimens and to determine whether the safety and tolerability profiles in healthy participants taking monthly doses of 600 mg or 800 mg tafenoquine are comparable in the same participants taking weekly 200 mg tafenoquine.

SECONDARY OUTCOMES:
Characterize the PK profiles of tafenoquine | six months
  A drug-free venous blood sample will be obtained from each participant at D0. PK blood sampling will be done to cover the absorption phase (Cabs, 1 to 4 hours after dosing), maximum concentration (Cmax, 22 to 24 hours after dosing), mid weekly or monthly concentration (Cmid) after dosing and the minimum concentration (Cmin) before the next dose of tafenoquine. PK parameters for each tafenoquine regimen will be calculated using a nonlinear mixed-effects modeling approach. The population PK model will evaluate the impact of clinically appropriate covariates, such as body weight, BMI, age and dose. Median (95% CI) Cmax and Cmin values of tafenoquine will also be estimated for the participants for each tafenoquine regimen.
Characterize the pharmacokinetic/pharmacodynamic (PK/PD) relationship | six months
  All collected PK samples will be analyzed using nonlinear mixed-effects modelling to describe the concentration-time profile of tafenoquine, and the association between drug exposure and potential adverse reactions. Different absorption and disposition models will be assessed to develop the structural PK model. Clinical covariates will be evaluated with a traditional forward addition/backward elimination approach, with particular focus on the influence of dose, body weight, BMI, and age. The PK model will be summarized by population mean estimates for structural model parameters, as well as estimated precision and between-patient variability in the same parameters. Secondary PK parameters, such as maximum and minimum tafenoquine concentrations, will be derived for each dosing regimen in order to evaluate the prospect of reaching effective concentrations for participants within each of the three tafenoquine regimens.
Determine the association of tafenoquine and its metabolite 5,6, orthoquinone in red blood cells | six months
  Because of the limited data on the association of tafenoquine in blood cells, venous blood and plasma samples will be measured in this study. Blood and plasma concentrations of tafenoquine and its metabolite, 5,6-orthoquinone will be quantified by liquid chromatography mass spectrometry (LCMS) in the selected reaction monitoring mode using heated electrospray ionization in positive ion mode. Blood and plasma samples (50 μL) will be precipitated with 200 μL of acetonitrile containing the internal standard. After centrifugation at 20,817 x g for 5 minutes at 4°C, an aliquot (10 μL) of the supernatant will be injected onto the analytical column.
  orthoquinone in red blood cells, the site of action of the drug's blood schizontocidal activity.
Determine the ex vivo antimalarial activity of tafenoquine in participants' plasma samples | six months
  Thirty participants will be invited to provide four additional 8 ml blood samples for assessing the ex vivo antimalarial activity of tafenoquine (TQ) and its metabolites. A blood sample will be collected before the 1st TQ dose to determine if their plasma can support the in vitro growth of P. falciparum isolates. After the collection of the pre-dose TQ blood sample, Cohort A participants will then provide additional blood samples after the 1st weekly 200 mg TQ dose and 1st monthly (600 mg and 800 mg) TQ doses. For Cohort B participants they will provide additional blood samples after the 2nd weekly 200 mg TQ dose and 2nd monthly (600 mg and 800 mg) TQ doses. Comparison of the inhibitory dilution of plasma samples on weekly and monthly TQ administration will be made to see which results in a 50% inhibition of uptake of [3H]-hypoxanthine (surrogate for parasite growth) compared to drugfree plasma samples (controls) against P. falciparum strains with different levels of drug.

CONTACTS AND LOCATIONS:
Overall Officials: Michael D Edstein, PhD, Principal Investigator — Australian Defence Force Malaria and Infectious Disease Institute
Locations (1):
- 108 Military Central Hospital, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No
All participants at the screening visit who fulfill the selection criteria and sign the ICF will be allocated a unique sequential screening study ID number by the clinical trial site. This will be a 3-digit number (starting at 001) prefixed by the letter "STQ" (i.e. STQ001, STQ002, etc. in ascending order). The letters "S" stands for screening and "TQ" for tafenoquine. A log of the screening ID numbers will be recorded in the register of data (RoD).

REFERENCES:
- [Background] Ackert J, Mohamed K, Slakter JS, El-Harazi S, Berni A, Gevorkyan H, Hardaker E, Hussaini A, Jones SW, Koh GCKW, Patel J, Rasmussen S, Kelly DS, Baranano DE, Thompson JT, Warren KA, Sergott RC, Tonkyn J, Wolstenholme A, Coleman H, Yuan A, Duparc S, Green JA. Randomized Placebo-Controlled Trial Evaluating the Ophthalmic Safety of Single-Dose Tafenoquine in Healthy Volunteers. Drug Saf. 2019 Sep;42(9):1103-1114. doi: 10.1007/s40264-019-00839-w. PMID 31187437
- [Background] Ashley EA, Pyae Phyo A, Woodrow CJ. Malaria. Lancet. 2018 Apr 21;391(10130):1608-1621. doi: 10.1016/S0140-6736(18)30324-6. Epub 2018 Apr 6. PMID 29631781
- [Background] Anh CX, Chavchich M, Birrell GW, Van Breda K, Travers T, Rowcliffe K, Lord AR, Shanks GD, Edstein MD. Pharmacokinetics and Ex Vivo Antimalarial Activity of Artesunate-Amodiaquine plus Methylene Blue in Healthy Volunteers. Antimicrob Agents Chemother. 2020 Feb 21;64(3):e01441-19. doi: 10.1128/AAC.01441-19. Print 2020 Feb 21. PMID 31907186
- [Background] Amato R, Pearson RD, Almagro-Garcia J, Amaratunga C, Lim P, Suon S, Sreng S, Drury E, Stalker J, Miotto O, Fairhurst RM, Kwiatkowski DP. Origins of the current outbreak of multidrug-resistant malaria in southeast Asia: a retrospective genetic study. Lancet Infect Dis. 2018 Mar;18(3):337-345. doi: 10.1016/S1473-3099(18)30068-9. Epub 2018 Feb 2. PMID 29398391
- [Background] Aronson NE, Sanders JW, Moran KA. In harm's way: infections in deployed American military forces. Clin Infect Dis. 2006 Oct 15;43(8):1045-51. doi: 10.1086/507539. Epub 2006 Sep 14. PMID 16983619
- [Background] Baird JK. Tafenoquine for travelers' malaria: evidence, rationale and recommendations. J Travel Med. 2018 Jan 1;25(1):tay110. doi: 10.1093/jtm/tay110. PMID 30380095
- [Background] Barrett O Jr, Skrzypek G, Datel W, Goldstein JD. Malaria imported to the United States from Vietnam. Chemoprophylaxis evaluated in returning soldiers. Am J Trop Med Hyg. 1969 Jul;18(4):495-9. doi: 10.4269/ajtmh.1969.18.495. No abstract available. PMID 5795444
- [Background] Battle KE, Lucas TCD, Nguyen M, Howes RE, Nandi AK, Twohig KA, Pfeffer DA, Cameron E, Rao PC, Casey D, Gibson HS, Rozier JA, Dalrymple U, Keddie SH, Collins EL, Harris JR, Guerra CA, Thorn MP, Bisanzio D, Fullman N, Huynh CK, Kulikoff X, Kutz MJ, Lopez AD, Mokdad AH, Naghavi M, Nguyen G, Shackelford KA, Vos T, Wang H, Lim SS, Murray CJL, Price RN, Baird JK, Smith DL, Bhatt S, Weiss DJ, Hay SI, Gething PW. Mapping the global endemicity and clinical burden of Plasmodium vivax, 2000-17: a spatial and temporal modelling study. Lancet. 2019 Jul 27;394(10195):332-343. doi: 10.1016/S0140-6736(19)31096-7. Epub 2019 Jun 19. PMID 31229233
- [Background] BECK AT, WARD CH, MENDELSON M, MOCK J, ERBAUGH J. An inventory for measuring depression. Arch Gen Psychiatry. 1961 Jun;4:561-71. doi: 10.1001/archpsyc.1961.01710120031004. No abstract available. PMID 13688369
- [Background] Beck HP, Wampfler R, Carter N, Koh G, Osorio L, Rueangweerayut R, Krudsood S, Lacerda MV, Llanos-Cuentas A, Duparc S, Rubio JP, Green JA. Estimation of the Antirelapse Efficacy of Tafenoquine, Using Plasmodium vivax Genotyping. J Infect Dis. 2016 Mar 1;213(5):794-9. doi: 10.1093/infdis/jiv508. Epub 2015 Oct 23. PMID 26500351
- [Background] Bellanger AP, Faucher JF, Robedat P, Schmitt A, Millon L, Hoen B. Malaria outbreak in French troops returning from Cote d'Ivoire. Scand J Infect Dis. 2011 Mar;43(3):230-3. doi: 10.3109/00365548.2010.538857. Epub 2010 Nov 25. PMID 21105845
- [Background] Bennett JW, Pybus BS, Yadava A, Tosh D, Sousa JC, McCarthy WF, Deye G, Melendez V, Ockenhouse CF. Primaquine failure and cytochrome P-450 2D6 in Plasmodium vivax malaria. N Engl J Med. 2013 Oct 3;369(14):1381-2. doi: 10.1056/NEJMc1301936. No abstract available. PMID 24088113
- [Background] Brisson M, Brisson P. Compliance with antimalaria chemoprophylaxis in a combat zone. Am J Trop Med Hyg. 2012 Apr;86(4):587-90. doi: 10.4269/ajtmh.2012.11-0511. PMID 22492140
- [Background] Charles BG, Miller AK, Nasveld PE, Reid MG, Harris IE, Edstein MD. Population pharmacokinetics of tafenoquine during malaria prophylaxis in healthy subjects. Antimicrob Agents Chemother. 2007 Aug;51(8):2709-15. doi: 10.1128/AAC.01183-06. Epub 2007 May 21. PMID 17517850
- [Background] Chu CS, Freedman DO. Tafenoquine and G6PD: a primer for clinicians. J Travel Med. 2019 Jun 1;26(4):taz023. doi: 10.1093/jtm/taz023. PMID 30941413
- [Background] Chua ACY, Ong JJY, Malleret B, Suwanarusk R, Kosaisavee V, Zeeman AM, Cooper CA, Tan KSW, Zhang R, Tan BH, Abas SN, Yip A, Elliot A, Joyner CJ, Cho JS, Breyer K, Baran S, Lange A, Maher SP, Nosten F, Bodenreider C, Yeung BKS, Mazier D, Galinski MR, Dereuddre-Bosquet N, Le Grand R, Kocken CHM, Renia L, Kyle DE, Diagana TT, Snounou G, Russell B, Bifani P. Robust continuous in vitro culture of the Plasmodium cynomolgi erythrocytic stages. Nat Commun. 2019 Aug 12;10(1):3635. doi: 10.1038/s41467-019-11332-4. PMID 31406175
- [Background] Coleman RE. Sporontocidal activity of the antimalarial WR-238605 against Plasmodium berghei ANKA in Anopheles stephensi. Am J Trop Med Hyg. 1990 Mar;42(3):196-205. doi: 10.4269/ajtmh.1990.42.196. PMID 2180334
- [Background] Coleman RE, Clavin AM, Milhous WK. Gametocytocidal and sporontocidal activity of antimalarials against Plasmodium berghei ANKA in ICR Mice and Anopheles stephensi mosquitoes. Am J Trop Med Hyg. 1992 Feb;46(2):169-82. doi: 10.4269/ajtmh.1992.46.169. PMID 1539752
- [Background] Commons RJ, McCarthy JS, Price RN. Tafenoquine for the radical cure and prevention of malaria: the importance of testing for G6PD deficiency. Med J Aust. 2020 Mar;212(4):152-153.e1. doi: 10.5694/mja2.50474. Epub 2020 Feb 9. No abstract available. PMID 32036613
- [Background] Daher A, Aljayyoussi G, Pereira D, Lacerda MVG, Alexandre MAA, Nascimento CT, Alves JC, da Fonseca LB, da Silva DMD, Pinto DP, Rodrigues DF, Silvino ACR, de Sousa TN, de Brito CFA, Ter Kuile FO, Lalloo DG. Pharmacokinetics/pharmacodynamics of chloroquine and artemisinin-based combination therapy with primaquine. Malar J. 2019 Sep 23;18(1):325. doi: 10.1186/s12936-019-2950-4. PMID 31547827
- [Background] Douglas AD, Baldeviano GC, Jin J, Miura K, Diouf A, Zenonos ZA, Ventocilla JA, Silk SE, Marshall JM, Alanine DGW, Wang C, Edwards NJ, Leiva KP, Gomez-Puerta LA, Lucas CM, Wright GJ, Long CA, Royal JM, Draper SJ. A defined mechanistic correlate of protection against Plasmodium falciparum malaria in non-human primates. Nat Commun. 2019 Apr 26;10(1):1953. doi: 10.1038/s41467-019-09894-4. PMID 31028254
- [Background] Dow GS, McCarthy WF, Reid M, Smith B, Tang D, Shanks GD. A retrospective analysis of the protective efficacy of tafenoquine and mefloquine as prophylactic anti-malarials in non-immune individuals during deployment to a malaria-endemic area. Malar J. 2014 Feb 6;13:49. doi: 10.1186/1475-2875-13-49. PMID 24502679
- [Background] Dow GS, Liu J, Lin G, Hetzell B, Thieling S, McCarthy WF, Tang D, Smith B. Summary of anti-malarial prophylactic efficacy of tafenoquine from three placebo-controlled studies of residents of malaria-endemic countries. Malar J. 2015 Nov 26;14:473. doi: 10.1186/s12936-015-0991-x. PMID 26610844
- [Background] Dow G, Smith B. The blood schizonticidal activity of tafenoquine makes an essential contribution to its prophylactic efficacy in nonimmune subjects at the intended dose (200 mg). Malar J. 2017 May 19;16(1):209. doi: 10.1186/s12936-017-1862-4. PMID 28526056
- [Background] Eastman RT, Fidock DA. Artemisinin-based combination therapies: a vital tool in efforts to eliminate malaria. Nat Rev Microbiol. 2009 Dec;7(12):864-74. doi: 10.1038/nrmicro2239. Epub 2009 Nov 2. PMID 19881520
- [Background] Ebstie YA, Abay SM, Tadesse WT, Ejigu DA. Tafenoquine and its potential in the treatment and relapse prevention of Plasmodium vivax malaria: the evidence to date. Drug Des Devel Ther. 2016 Jul 26;10:2387-99. doi: 10.2147/DDDT.S61443. eCollection 2016. PMID 27528800
- [Background] Edstein MD, Kocisko DA, Brewer TG, Walsh DS, Eamsila C, Charles BG. Population pharmacokinetics of the new antimalarial agent tafenoquine in Thai soldiers. Br J Clin Pharmacol. 2001 Dec;52(6):663-70. doi: 10.1046/j.0306-5251.2001.01482.x. PMID 11736877
- [Background] Edstein MD, Kocisko DA, Walsh DS, Eamsila C, Charles BG, Rieckmann KH. Plasma concentrations of tafenoquine, a new long-acting antimalarial agent, in thai soldiers receiving monthly prophylaxis. Clin Infect Dis. 2003 Dec 15;37(12):1654-8. doi: 10.1086/379718. Epub 2003 Nov 20. PMID 14689348
- [Background] Eick-Cost AA, Hu Z, Rohrbeck P, Clark LL. Neuropsychiatric Outcomes After Mefloquine Exposure Among U.S. Military Service Members. Am J Trop Med Hyg. 2017 Jan 11;96(1):159-166. doi: 10.4269/ajtmh.16-0390. Epub 2016 Nov 14. PMID 28077744
- [Background] Elmes NJ, Nasveld PE, Kitchener SJ, Kocisko DA, Edstein MD. The efficacy and tolerability of three different regimens of tafenoquine versus primaquine for post-exposure prophylaxis of Plasmodium vivax malaria in the Southwest Pacific. Trans R Soc Trop Med Hyg. 2008 Nov;102(11):1095-101. doi: 10.1016/j.trstmh.2008.04.024. Epub 2008 Jun 9. PMID 18541280
- [Background] Fernando SD, Ranaweera D, Weerasena MS, Booso R, Wickramasekara T, Madurapperuma CP, Danansuriya M, Rodrigo C, Herath H. Success of malaria chemoprophylaxis for outbound civil and military travellers in prevention of reintroduction of malaria in Sri Lanka. Int Health. 2020 Jul 1;12(4):332-338. doi: 10.1093/inthealth/ihz094. PMID 31927579
- [Background] Frampton JE. Tafenoquine: First Global Approval. Drugs. 2018 Sep;78(14):1517-1523. doi: 10.1007/s40265-018-0979-2. PMID 30229442
- [Background] Fry M, Pudney M. Site of action of the antimalarial hydroxynaphthoquinone, 2-[trans-4-(4'-chlorophenyl) cyclohexyl]-3-hydroxy-1,4-naphthoquinone (566C80). Biochem Pharmacol. 1992 Apr 1;43(7):1545-53. doi: 10.1016/0006-2952(92)90213-3. PMID 1314606
- [Background] Fukuda MM, Krudsood S, Mohamed K, Green JA, Warrasak S, Noedl H, Euswas A, Ittiverakul M, Buathong N, Sriwichai S, Miller RS, Ohrt C. A randomized, double-blind, active-control trial to evaluate the efficacy and safety of a three day course of tafenoquine monotherapy for the treatment of Plasmodium vivax malaria. PLoS One. 2017 Nov 9;12(11):e0187376. doi: 10.1371/journal.pone.0187376. eCollection 2017. PMID 29121061
- [Background] Fukuda MM, Wojnarski M, Martin N, Zottig V, Waters NC. Editorial: Malaria in the Korean peninsula: Risk factors, latent infections, and the possible role of tafenoquine, a new antimalarial weapon. MSMR. 2018 Nov;25(11):2-3. No abstract available. PMID 30475635
- [Background] Green JA, Patel AK, Patel BR, Hussaini A, Harrell EJ, McDonald MJ, Carter N, Mohamed K, Duparc S, Miller AK. Tafenoquine at therapeutic concentrations does not prolong Fridericia-corrected QT interval in healthy subjects. J Clin Pharmacol. 2014 Sep;54(9):995-1005. doi: 10.1002/jcph.302. Epub 2014 Apr 9. PMID 24700490
- [Background] Hale BR, Owusu-Agyei S, Fryauff DJ, Koram KA, Adjuik M, Oduro AR, Prescott WR, Baird JK, Nkrumah F, Ritchie TL, Franke ED, Binka FN, Horton J, Hoffman SL. A randomized, double-blind, placebo-controlled, dose-ranging trial of tafenoquine for weekly prophylaxis against Plasmodium falciparum. Clin Infect Dis. 2003 Mar 1;36(5):541-9. doi: 10.1086/367542. Epub 2003 Feb 14. PMID 12594633
- [Background] Hamilton WL, Amato R, van der Pluijm RW, Jacob CG, Quang HH, Thuy-Nhien NT, Hien TT, Hongvanthong B, Chindavongsa K, Mayxay M, Huy R, Leang R, Huch C, Dysoley L, Amaratunga C, Suon S, Fairhurst RM, Tripura R, Peto TJ, Sovann Y, Jittamala P, Hanboonkunupakarn B, Pukrittayakamee S, Chau NH, Imwong M, Dhorda M, Vongpromek R, Chan XHS, Maude RJ, Pearson RD, Nguyen T, Rockett K, Drury E, Goncalves S, White NJ, Day NP, Kwiatkowski DP, Dondorp AM, Miotto O. Evolution and expansion of multidrug-resistant malaria in southeast Asia: a genomic epidemiology study. Lancet Infect Dis. 2019 Sep;19(9):943-951. doi: 10.1016/S1473-3099(19)30392-5. Epub 2019 Jul 22. PMID 31345709
- [Background] Happi CT, Gbotosho GO, Folarin OA, Milner D, Sarr O, Sowunmi A, Kyle DE, Milhous WK, Wirth DF, Oduola AM. Confirmation of emergence of mutations associated with atovaquone-proguanil resistance in unexposed Plasmodium falciparum isolates from Africa. Malar J. 2006 Oct 4;5:82. doi: 10.1186/1475-2875-5-82. PMID 17020611
- [Background] Hounkpatin AB, Kreidenweiss A, Held J. Clinical utility of tafenoquine in the prevention of relapse of Plasmodium vivax malaria: a review on the mode of action and emerging trial data. Infect Drug Resist. 2019 Mar 6;12:553-570. doi: 10.2147/IDR.S151031. eCollection 2019. PMID 30881061
- [Background] Klein TA, Seyoum B, Forshey BM, Ellis KK, McCall H, Jackson K, Tucker C, Yi S, Kim M, Kim H. Cluster of vivax malaria in U.S. soldiers training near the demilitarized zone, Republic of Korea during 2015. MSMR. 2018 Nov;25(11):4-9. PMID 30475636
- [Background] Korsinczky M, Chen N, Kotecka B, Saul A, Rieckmann K, Cheng Q. Mutations in Plasmodium falciparum cytochrome b that are associated with atovaquone resistance are located at a putative drug-binding site. Antimicrob Agents Chemother. 2000 Aug;44(8):2100-8. doi: 10.1128/AAC.44.8.2100-2108.2000. PMID 10898682
- [Background] Lacerda MVG, Llanos-Cuentas A, Krudsood S, Lon C, Saunders DL, Mohammed R, Yilma D, Batista Pereira D, Espino FEJ, Mia RZ, Chuquiyauri R, Val F, Casapia M, Monteiro WM, Brito MAM, Costa MRF, Buathong N, Noedl H, Diro E, Getie S, Wubie KM, Abdissa A, Zeynudin A, Abebe C, Tada MS, Brand F, Beck HP, Angus B, Duparc S, Kleim JP, Kellam LM, Rousell VM, Jones SW, Hardaker E, Mohamed K, Clover DD, Fletcher K, Breton JJ, Ugwuegbulam CO, Green JA, Koh GCKW. Single-Dose Tafenoquine to Prevent Relapse of Plasmodium vivax Malaria. N Engl J Med. 2019 Jan 17;380(3):215-228. doi: 10.1056/NEJMoa1710775. PMID 30650322
- [Background] Lalani T, Yun H, Tribble D, Ganesan A, Kunz A, Fairchok M, Schnaubelt E, Fraser J, Mitra I, Kronmann KC, Burgess T, Deiss RG, Riddle MS, Johnson MD. A comparison of compliance rates with anti-vectorial protective measures during travel to regions with dengue or chikungunya activity, and regions endemic for Plasmodium falciparum malaria. J Travel Med. 2016 Jul 4;23(5):taw043. doi: 10.1093/jtm/taw043. Print 2016 May. PMID 27378367
- [Background] Landman KZ, Tan KR, Arguin PM. Adherence to malaria prophylaxis among Peace Corps Volunteers in the Africa region, 2013. Travel Med Infect Dis. 2015 Jan-Feb;13(1):61-8. doi: 10.1016/j.tmaid.2014.12.001. Epub 2014 Dec 11. PMID 25534297
- [Background] Llanos-Cuentas A, Lacerda MV, Rueangweerayut R, Krudsood S, Gupta SK, Kochar SK, Arthur P, Chuenchom N, Mohrle JJ, Duparc S, Ugwuegbulam C, Kleim JP, Carter N, Green JA, Kellam L. Tafenoquine plus chloroquine for the treatment and relapse prevention of Plasmodium vivax malaria (DETECTIVE): a multicentre, double-blind, randomised, phase 2b dose-selection study. Lancet. 2014 Mar 22;383(9922):1049-58. doi: 10.1016/S0140-6736(13)62568-4. Epub 2013 Dec 19. PMID 24360369
- [Background] Llanos-Cuentas A, Lacerda MVG, Hien TT, Velez ID, Namaik-Larp C, Chu CS, Villegas MF, Val F, Monteiro WM, Brito MAM, Costa MRF, Chuquiyauri R, Casapia M, Nguyen CH, Aruachan S, Papwijitsil R, Nosten FH, Bancone G, Angus B, Duparc S, Craig G, Rousell VM, Jones SW, Hardaker E, Clover DD, Kendall L, Mohamed K, Koh GCKW, Wilches VM, Breton JJ, Green JA. Tafenoquine versus Primaquine to Prevent Relapse of Plasmodium vivax Malaria. N Engl J Med. 2019 Jan 17;380(3):229-241. doi: 10.1056/NEJMoa1802537. PMID 30650326
- [Background] Lourens C, Lindegardh N, Barnes KI, Guerin PJ, Sibley CH, White NJ, Tarning J. Benefits of a pharmacology antimalarial reference standard and proficiency testing program provided by the Worldwide Antimalarial Resistance Network (WWARN). Antimicrob Agents Chemother. 2014 Jul;58(7):3889-94. doi: 10.1128/AAC.02362-14. Epub 2014 Apr 28. PMID 24777099
- [Background] McCarthy JS, Smith B, Reid M, Berman J, Marquart L, Dobbin C, West L, Read LT, Dow GS. Blood Schizonticidal Activity and Safety of Tafenoquine When Administered as Chemoprophylaxis to Healthy, Nonimmune Participants Followed by Blood Stage Plasmodium falciparum Challenge: A Randomized, Double-blind, Placebo-controlled Phase 1b Study. Clin Infect Dis. 2019 Jul 18;69(3):480-486. doi: 10.1093/cid/ciy939. PMID 30388194
- [Background] Nasveld P, Kitchener S. Treatment of acute vivax malaria with tafenoquine. Trans R Soc Trop Med Hyg. 2005 Jan;99(1):2-5. doi: 10.1016/j.trstmh.2004.01.013. PMID 15550254
- [Background] Nasveld PE, Edstein MD, Reid M, Brennan L, Harris IE, Kitchener SJ, Leggat PA, Pickford P, Kerr C, Ohrt C, Prescott W; Tafenoquine Study Team. Randomized, double-blind study of the safety, tolerability, and efficacy of tafenoquine versus mefloquine for malaria prophylaxis in nonimmune subjects. Antimicrob Agents Chemother. 2010 Feb;54(2):792-8. doi: 10.1128/AAC.00354-09. Epub 2009 Dec 7. PMID 19995933
- [Background] Newton JA Jr, Schnepf GA, Wallace MR, Lobel HO, Kennedy CA, Oldfield EC 3rd. Malaria in US Marines returning from Somalia. JAMA. 1994 Aug 3;272(5):397-9. PMID 8028173
- [Background] Nicolas B, Papillault des Charbonnieres L, Vasseur T, Mauclere P. Assessment of adherence to malaria chemoprophylaxis in a French Navy frigate deployed in Southeast Asia. Med Sante Trop. 2017 Jun 1;27(2):155-159. doi: 10.1684/mst.2017.0666. PMID 28572077
- [Background] Novitt-Moreno A, Ransom J, Dow G, Smith B, Read LT, Toovey S. Tafenoquine for malaria prophylaxis in adults: An integrated safety analysis. Travel Med Infect Dis. 2017 May-Jun;17:19-27. doi: 10.1016/j.tmaid.2017.05.008. Epub 2017 May 8. PMID 28495354
- [Background] Pang LW, Limsomwong N, Boudreau EF, Singharaj P. Doxycycline prophylaxis for falciparum malaria. Lancet. 1987 May 23;1(8543):1161-4. doi: 10.1016/s0140-6736(87)92141-6. PMID 2883488
- [Background] Petersen E. The safety of atovaquone/proguanil in long-term malaria prophylaxis of nonimmune adults. J Travel Med. 2003 May;10 Suppl 1:S13-5; discussion S21. doi: 10.2310/7060.2003.35050. PMID 12737755
- [Background] Plucinski MM, Huber CS, Akinyi S, Dalton W, Eschete M, Grady K, Silva-Flannery L, Mathison BA, Udhayakumar V, Arguin PM, Barnwell JW. Novel Mutation in Cytochrome B of Plasmodium falciparum in One of Two Atovaquone-Proguanil Treatment Failures in Travelers Returning From Same Site in Nigeria. Open Forum Infect Dis. 2014 Aug 5;1(2):ofu059. doi: 10.1093/ofid/ofu059. eCollection 2014 Sep. PMID 25734129
- [Background] Ponsa N, Sattabongkot J, Kittayapong P, Eikarat N, Coleman RE. Transmission-blocking activity of tafenoquine (WR-238605) and artelinic acid against naturally circulating strains of Plasmodium vivax in Thailand. Am J Trop Med Hyg. 2003 Nov;69(5):542-7. PMID 14695093
- [Background] Quang NN, Chavchich M, Anh CX, Birrell GW, van Breda K, Travers T, Rowcliffe K, Edstein MD. Comparison of the Pharmacokinetics and Ex Vivo Antimalarial Activities of Artesunate-Amodiaquine and Artemisinin-Piperaquine in Healthy Volunteers for Preselection Malaria Therapy. Am J Trop Med Hyg. 2018 Jul;99(1):65-72. doi: 10.4269/ajtmh.17-0434. Epub 2018 May 3. PMID 29741150
- [Background] Rogers WO, Sem R, Tero T, Chim P, Lim P, Muth S, Socheat D, Ariey F, Wongsrichanalai C. Failure of artesunate-mefloquine combination therapy for uncomplicated Plasmodium falciparum malaria in southern Cambodia. Malar J. 2009 Jan 12;8:10. doi: 10.1186/1475-2875-8-10. PMID 19138388
- [Background] Rutherford AE, Yale RS, Finn MF. Malaria Prophylaxis Adherence Among Aircrew Members. Aerosp Med Hum Perform. 2019 Jul 1;90(7):643-646. doi: 10.3357/AMHP.5306.2019. PMID 31227039
- [Background] Saunders D, Duplessis C, Lescano A, Andagalu B, Thomas A, Fukuda M, Cummings J; US DoD Malaria Surveillance Investigators Group. US Department of Defense contributions to malaria surveillance. Lancet Infect Dis. 2013 Apr;13(4):293-4. doi: 10.1016/S1473-3099(13)70065-3. No abstract available. PMID 23538221
- [Background] Saunders DL, Garges E, Manning JE, Bennett K, Schaffer S, Kosmowski AJ, Magill AJ. Safety, Tolerability, and Compliance with Long-Term Antimalarial Chemoprophylaxis in American Soldiers in Afghanistan. Am J Trop Med Hyg. 2015 Sep;93(3):584-90. doi: 10.4269/ajtmh.15-0245. Epub 2015 Jun 29. PMID 26123954
- [Background] Schneiderman AI, Cypel YS, Dursa EK, Bossarte RM. Associations between Use of Antimalarial Medications and Health among U.S. Veterans of the Wars in Iraq and Afghanistan. Am J Trop Med Hyg. 2018 Sep;99(3):638-648. doi: 10.4269/ajtmh.18-0107. Epub 2018 Jun 21. PMID 29943726
- [Background] Schwartz E. Prophylaxis of malaria. Mediterr J Hematol Infect Dis. 2012;4(1):e2012045. doi: 10.4084/MJHID.2012.45. Epub 2012 Jun 29. PMID 22811794
- [Background] Shah NK, Alker AP, Sem R, Susanti AI, Muth S, Maguire JD, Duong S, Ariey F, Meshnick SR, Wongsrichanalai C. Molecular surveillance for multidrug-resistant Plasmodium falciparum, Cambodia. Emerg Infect Dis. 2008 Oct;14(10):1637-40. doi: 10.3201/eid1410.080080. PMID 18826834
- [Background] Shanks GD, Oloo AJ, Aleman GM, Ohrt C, Klotz FW, Braitman D, Horton J, Brueckner R. A new primaquine analogue, tafenoquine (WR 238605), for prophylaxis against Plasmodium falciparum malaria. Clin Infect Dis. 2001 Dec 15;33(12):1968-74. doi: 10.1086/324081. Epub 2001 Nov 7. PMID 11700577
- [Background] Spring MD, Sousa JC, Li Q, Darko CA, Morrison MN, Marcsisin SR, Mills KT, Potter BM, Paolino KM, Twomey PS, Moon JE, Tosh DM, Cicatelli SB, Froude JW, Pybus BS, Oliver TG, McCarthy WF, Waters NC, Smith PL, Reichard GA, Bennett JW. Determination of Cytochrome P450 Isoenzyme 2D6 (CYP2D6) Genotypes and Pharmacogenomic Impact on Primaquine Metabolism in an Active-Duty US Military Population. J Infect Dis. 2019 Oct 22;220(11):1761-1770. doi: 10.1093/infdis/jiz386. PMID 31549155
- [Background] St Jean PL, Xue Z, Carter N, Koh GC, Duparc S, Taylor M, Beaumont C, Llanos-Cuentas A, Rueangweerayut R, Krudsood S, Green JA, Rubio JP. Tafenoquine treatment of Plasmodium vivax malaria: suggestive evidence that CYP2D6 reduced metabolism is not associated with relapse in the Phase 2b DETECTIVE trial. Malar J. 2016 Feb 18;15:97. doi: 10.1186/s12936-016-1145-5. PMID 26888075
- [Background] Terrell AG, Forde ME, Firth R, Ross DA. Malaria Chemoprophylaxis and Self-Reported Impact on Ability to Work: Mefloquine Versus Doxycycline. J Travel Med. 2015 Nov-Dec;22(6):383-8. doi: 10.1111/jtm.12232. Epub 2015 Oct 1. PMID 26424621
- [Background] Thakkar N, Green JA, Koh GCKW, Duparc S, Tenero D, Goyal N. Population Pharmacokinetics of Tafenoquine, a Novel Antimalarial. Antimicrob Agents Chemother. 2018 Oct 24;62(11):e00711-18. doi: 10.1128/AAC.00711-18. Print 2018 Nov. PMID 30201820
- [Background] Vinayak S, Alam MT, Sem R, Shah NK, Susanti AI, Lim P, Muth S, Maguire JD, Rogers WO, Fandeur T, Barnwell JW, Escalante AA, Wongsrichanalai C, Ariey F, Meshnick SR, Udhayakumar V. Multiple genetic backgrounds of the amplified Plasmodium falciparum multidrug resistance (pfmdr1) gene and selective sweep of 184F mutation in Cambodia. J Infect Dis. 2010 May 15;201(10):1551-60. doi: 10.1086/651949. PMID 20367478
- [Background] Walsh DS, Looareesuwan S, Wilairatana P, Heppner DG Jr, Tang DB, Brewer TG, Chokejindachai W, Viriyavejakul P, Kyle DE, Milhous WK, Schuster BG, Horton J, Braitman DJ, Brueckner RP. Randomized dose-ranging study of the safety and efficacy of WR 238605 (Tafenoquine) in the prevention of relapse of Plasmodium vivax malaria in Thailand. J Infect Dis. 1999 Oct;180(4):1282-7. doi: 10.1086/315034. PMID 10479159
- [Background] Walsh DS, Wilairatana P, Tang DB, Heppner DG Jr, Brewer TG, Krudsood S, Silachamroon U, Phumratanaprapin W, Siriyanonda D, Looareesuwan S. Randomized trial of 3-dose regimens of tafenoquine (WR238605) versus low-dose primaquine for preventing Plasmodium vivax malaria relapse. Clin Infect Dis. 2004 Oct 15;39(8):1095-103. doi: 10.1086/424508. Epub 2004 Sep 24. PMID 15486831
- [Background] Walsh DS, Eamsila C, Sasiprapha T, Sangkharomya S, Khaewsathien P, Supakalin P, Tang DB, Jarasrumgsichol P, Cherdchu C, Edstein MD, Rieckmann KH, Brewer TG. Efficacy of monthly tafenoquine for prophylaxis of Plasmodium vivax and multidrug-resistant P. falciparum malaria. J Infect Dis. 2004 Oct 15;190(8):1456-63. doi: 10.1086/424468. Epub 2004 Sep 20. PMID 15378438
- [Background] Warrasak S, Euswas A, Fukuda MM, Ittiverakul M, Miller RS, Krudsood S, Ohrt C. Comparative ophthalmic assessment of patients receiving tafenoquine or chloroquine/primaquine in a randomized clinical trial for Plasmodium vivax malaria radical cure. Int Ophthalmol. 2019 Aug;39(8):1767-1782. doi: 10.1007/s10792-018-1003-2. Epub 2018 Sep 29. PMID 30269312
- [Background] Wellems TE, Plowe CV. Chloroquine-resistant malaria. J Infect Dis. 2001 Sep 15;184(6):770-6. doi: 10.1086/322858. Epub 2001 Aug 7. PMID 11517439
- [Background] Whitman TJ, Coyne PE, Magill AJ, Blazes DL, Green MD, Milhous WK, Burgess TH, Freilich D, Tasker SA, Azar RG, Endy TP, Clagett CD, Deye GA, Shanks GD, Martin GJ. An outbreak of Plasmodium falciparum malaria in U.S. Marines deployed to Liberia. Am J Trop Med Hyg. 2010 Aug;83(2):258-65. doi: 10.4269/ajtmh.2010.09-0774. PMID 20682864
- [Background] Woodrow CJ, White NJ. The clinical impact of artemisinin resistance in Southeast Asia and the potential for future spread. FEMS Microbiol Rev. 2017 Jan;41(1):34-48. doi: 10.1093/femsre/fuw037. Epub 2016 Sep 8. PMID 27613271
- [Background] Wojnarski M, Lon C, Vanachayangkul P, Gosi P, Sok S, Rachmat A, Harrison D, Berjohn CM, Spring M, Chaoratanakawee S, Ittiverakul M, Buathong N, Chann S, Wongarunkochakorn S, Waltmann A, Kuntawunginn W, Fukuda MM, Burkly H, Heang V, Heng TK, Kong N, Boonchan T, Chum B, Smith P, Vaughn A, Prom S, Lin J, Lek D, Saunders D. Atovaquone-Proguanil in Combination With Artesunate to Treat Multidrug-Resistant P. falciparum Malaria in Cambodia: An Open-Label Randomized Trial. Open Forum Infect Dis. 2019 Sep 4;6(9):ofz314. doi: 10.1093/ofid/ofz314. eCollection 2019 Sep. PMID 31660398
- See also: World Health Organization Malaria Report 2019 — https://www.who.int/malaria/publications/world-malaria-report-2019/en/
- See also: Tafenoquine (Arakoda) U.S. prescribing information 2018 — https://www.accessdata.fda.gov/drugsatfda_docs/label/2018/210607lbl.pdf
- See also: Tafenoquine approval for Australia — https://e69f947d-9273-4db6-8a44689a919a5ca4.filesusr.com/ugd/d8a71c_107482fde91046b9af73cc5b3b9c117b.pdf
- See also: ICMJE Defining Roles of Authors and Contributors — http://www.icmje.org/recommendations/browse/roles-and-responsibilities/defining-the-role-of-authors-and-contributors.html
- See also: U.S. FDA Tafenoquine (Krintafel) — https://www.accessdata.fda.gov/drugsatfda_docs/nda/2018/210795Orig1s000TOC.cfm
- See also: U.S. FDA Guidance on Drug Induced Liver Injury: Premarketing Clinical Evaluation 2009 — https://www.fda.gov/media/116737/download
- See also: Arakoda package insert — https://www.accessdata.fda.gov/drugsatfda_docs/label/2018/210607lbl.pdf